CLINICAL TRIAL: NCT06184087
Title: Childbirth Education on Upright Positions and Mobility During Labor
Brief Title: Childbirth Education on Upright Positions Mobility During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Hana Borrer (Unknown)
Responsible Party: Principal Investigator, Ilana Dubovi, Senior Lecturer, Tel Aviv University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TelAvivU_Childbirth education
Record Dates: First submitted 2023-12-04; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Childbirth Classes
Keywords: childbirth education; upright positions; mobility during labor

STUDY DESIGN:
Intervention Model Description: A prospective quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): The control group (n = 34) participated in routine childbirth education. The group received the same content via a childbirth class as the intervention group of five meetings (a total of 12.5 hours) given by a nurse midwife.
  Women in the control group received a routine instructional approach which was based on lectures, videos, discussions, and practice/rehearsals.
  Interventions: Other: Educational/Instructional
- Intervention group (Experimental): The intervention group (n= 36) learned with childbirth education that included interactive and constructive cognitive engagement activities.
  The intervention group received the same content as the control group (a total of 12.5 hours), however, the content regarding upright positions and mobility was instructed using the ICAP constructive-interactive engagement modes.
  Interventions: Other: Educational/Instructional

INTERVENTIONS:
Other: Educational/Instructional — ICAP constructive-interactive engagement mode

SUMMARY:
Background and study aims: A prospective quasi-experimental study will be conducted among nulliparous women from the ultra-orthodox Jewish community.

Study design: While the control group participated in routine childbirth education, the intervention group learned with childbirth education that included interactive and constructive cognitive engagement activities. Participants in both groups completed a set of questionnaires regarding knowledge, attitudes, and self-efficacy.

DETAILED DESCRIPTION:
Background: Upright labor positions and movement during labor have a positive effect on childbirth, yet the predominant labor positions are still horizontal. Therefore, it is important to explore how it is possible to improve childbirth education, particularly its instructional design, to strengthen women's self-efficacy toward the use of upright positions and mobility during labor. The aim of the study was to evaluate the impact of an instructional approach based on a cognitive engagement ICAP (Interactive, Constructive, Active, Passive) framework on the development of knowledge, attitudes, and self-efficacy expectations toward upright positions and mobility during labor.

Methods: A prospective quasi-experimental study was conducted among nulliparous women from the ultra-orthodox Jewish community (n=74). While the control group (n = 34) participated in routine childbirth education, the intervention group (n = 36) learned with childbirth education that included interactive and constructive cognitive engagement activities. Participants in both groups completed a set of questionnaires regarding knowledge, attitudes, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women

Exclusion Criteria:

*High-risk pregnancy

Max Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The study is about nulliparous women labor class
Enrollment: 74 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Self-efficacy toward upright positions and mobility during labor | The questionnaire was administered at the beginning of the childbirth course and again at the end of the fifth meeting of the childbirth course.
  The Childbirth Self-Efficacy Inventory that was developed by Lowe (2000).The participants were asked to rank on a 1-10 Likert scale 18 listed behaviors for how much they can help to cope with labor.

SECONDARY OUTCOMES:
Attitudes towards upright positions and mobility during labor | The questionnaire was administered at the beginning of the childbirth course and again at the end of the fifth meeting of the childbirth course.
  Questionnaire that was constructed according to Ajzen (1991) which defines attitudes as the positive or negative evaluation of certain behavior. The questionnaire includes 6 items; the participants are asked to rank their attitudes on a seven-point Osgood differential semantic scale, where 1 represents negative attitudes, and 7 represents positive attitudes. Higher score means a stronger attitude toward upright positions and mobility during labor.
Knowledge about positions and mobility during labor | The questionnaire was administered at the beginning of the childbirth course and again at the end of the fifth meeting of the childbirth course.
  Knowledge questionnaire about labor positions and mobility was developed and validated by the authors.

CONTACTS AND LOCATIONS:
Locations (1):
- Merkaz Shifra, Modi'in Illit, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Will be provided upon request